CLINICAL TRIAL: NCT03532113
Title: Memory and Cognitive Control for Optimal Aging: Study on the Effect of Cognitive Interventions, Cerebral Mechanisms Involved and Processes Promoting Transfer
Brief Title: Attentional Control Training in Older Adults: Efficacy, Transfer and Brain Substrates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Sylvie Belleville, Research director of CRIUGM and full professor at University of Montreal, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRIUGM-005
Record Dates: First submitted 2018-04-18; First posted 2018-05-22 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Inhibition (Psychology); Updating; General Knowledge; No Training
Keywords: Cognitive intervention; Cognitive training; Aging; Working memory; Cognitive reserve; Brain imaging; Brain plasticity; Polymorphisms; Transfer; Inhibition; Updating
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Older participants are randomly assigned to one of three intervention conditions (Inhibition ; Updating ; General knowledge).
  Young participants only complete the initial assessment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The experimenters are blind in the clinical trials. Participants know that there are different training programs but they ignore the purpose of each one.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Updating (Experimental): The Updating intervention aims to improve the ability to monitor and quickly add or delete of content of working memory.
  Interventions: Behavioral: Updating
- Inhibition (Experimental): The Inhibition intervention aims to improve the ability to supersede responses that are prepotent or automatic for a given situation.
  Interventions: Behavioral: Inhibition
- General Knowledge (Active Comparator): The General knowledge intervention allows the learning of information on various topics. It does not involve attentional control but semantic knowledge.
  Interventions: Behavioral: General knowledge

INTERVENTIONS:
Behavioral: Updating — Updating is trained across 12 sessions using N-back-type exercises. Training is performed on a samsung galaxy tab2. Each session lasts 30 minutes. The difficult is reset and the nature of the stimuli (numbers vs. symbols) is changed halfway in each session.
  Arms: Updating
Behavioral: Inhibition — Inhibition is trained across 12 sessions with Stroop-like exercises. Training is performed on a samsung galaxy tab2. Each session lasts 30 minutes. The difficult is reset and the nature of stimuli (letters vs. numbers) is changed halfway in each session.
  Arms: Inhibition
Behavioral: General knowledge — General Knowledge is trained across 12 sessions. Participants complete four-choice questions relating to general knowledge and vocabulary and are provided with the correct answer and a short explanation. Questions are displayed one by one on a computer screen with a maximum of 20 seconds per question. Each session lasts 30 minutes and includes 2 blocks of 40 new questions each (about 220 seconds per block). Questions with wrong answers are displayed again at the end of each block.
  Arms: General Knowledge

SUMMARY:
Formal education and cognitively stimulating hobbies and profession have a protective effect against age-related cognitive decline and Alzheimer's disease. It is therefore possible that providing cognitively stimulating interventions at a later age increases neuroplasticity and brain resilience. Processes of updating and inhibition are both impaired by aging. Several studies have shown that updating can be improved but very few studies targeted inhibition in spite of the fact that it is impaired in older adults. The aim of this study is to assess the effect of cognitive interventions that will target either of these two components. The investigators will examine the effect on behavior, brain measures and transfer tasks. The investigators will also assess whether the efficacy varies as a function of personal variables such as prior cognitive profile, reserve proxies, genetic polymorphisms and brain markers.

DETAILED DESCRIPTION:
Formal education and cognitively stimulating hobbies and profession have a protective effect against age-related cognitive decline and Alzheimer's disease. The cognitive reserve model suggests that engaging in cognitively stimulating activities may induce brain processes and/or morphological characteristics that make individuals more resilient to the effects of brain damage. It is therefore possible that providing cognitive interventions at a later age amplify similar neuroplastic processes and thus reduce the deleterious effects of aging. Cognitive interventions refer to programs and/or strategies aimed at increasing or optimizing cognitive performance. Many of these programs target working memory (WM), which is defined as the ability to control attention in order to keep information active and accessible. Miyake's influential model proposes that WM relies on the coordinated functioning of a small set of attentional control components. Here the investigators will focus on two of these components: inhibition and updating. Training those two components might reveal critical as they are impaired in aging and subtend a range of more complex cognitive processes. Furthermore, they rely on distinct brain networks and are sensitive to cognitive lifestyle. Several studies have shown that updating capacities of older adults can be improved by cognitive training but very few studies targeted inhibition in spite of the fact that it is severly impaired by aging. The aim of this study is to assess the effect of cognitive interventions that will target either of these two components and compare their effect to that of an active control training. The investigators will examine their effect on behavior, brain measures and transfer tasks. The investigators will also assess whether the efficacy varies as a function of personal variables such as prior cognitive profile, reserve proxies, genetic polymorphisms and brain markers. The investigators will also examine the cumulative effect of training by measuring efficacy at three time points for the proximal outcomes and at five time points for the distal outcomes. Finally, a group of younger adults will be tested at baseline to assess whether training normalize performance, that is, whether the performance of older adults after training is improved to the level of typical young adults.

90 healthy older adults (60-85 years) will be recruited for this study, as well as thirty young adults (20-35 years) who will complete only the initial assessment (PRE). All participants will be recruited from the community and living in the Montreal area. A telephone interview will provide initial selection information. Eligible persons will be invited to come to the laboratory for a standardized clinical and neuropsychological battery in order to evaluate their clinical status and cognitive functioning. The older adults will be randomly assigned to one of three intervention conditions (Inhibition, Updating, Active control). Updating will be trained using N-back-like exercises whereas inhibition will be trained with Stroop-like exercises. Different types of stimuli will be used to facilitate transfer. The control intervention will include exercises on general knowledge and vocabulary. All training will be computerized. Training will be provided in 12 half-hours training sessions. Outcome measures will be taken no more than two weeks prior to training (PRE), between Session 6 and 7 (POST1) and no more than one week following Session 12 (POST2). Participants will be trained in small groups of 6 to 10 individuals recruited in about 6 waves. The first two waves will allow to pilot the procedure/team and will be accrued to the whole trial if the training procedure and outcome measures remain unchanged.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking
* Right-handed
* Sufficient visual and auditory acuity to undergo neuropsychological tests and to do the interventions.
* Sufficient delayed recall score above the education-adjusted cut-offs (≥9 for 16+ years of education; ≥5 for 8-15 years of education; ≥3 for 0-7 years of education) at the Logical Memory test (Wechsler Memory Scale, maximum score 25).

Exclusion Criteria:

* Answer 'Yes' to the two following questions: "Do you feel like your memory is becoming worse?" "Does this worry you?" (to exclude subjective cognitive decline).
* The presence of a disease or injury of the central nervous system: moderate to severe chronic static leukoencephalopathy (including previous traumatic injury), multiple sclerosis, a serious developmental handicap, subdural hematoma (past or current), subarachnoid haemorrhage (past or current), primary cerebral tumour or cerebral metastases, epilepsy (current), dementia or another neurodegenerative disease, and other rarer brain illnesses.
* Symptomatic stroke within the previous year.
* Alcoholism or substance abuse
* History of intracranial surgery.
* Major surgery within last 2 months.
* General anesthesia in the past 6 months.
* Serious comorbid condition that, in the opinion of the study investigator, is likely to result in death within a year.
* Major depression or anxiety.
* Schizophrenia or other major psychiatric disorder (e.g., bipolar disorder).
* Individuals where French is not sufficiently proficient for clinical assessment and neuropsychological testing.
* Unable to undergo MRI scan due to medical contraindications or inability to tolerate the procedure.
* Plans on moving outside the province within the next 2 months.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Changes on the updating composite measure (Proximal outcome). | within the 2 weeks before intervention starts; 3rd week after intervention starts (after the 6th training session); 6th week (after the 12th training session)
  An updating composite score will be computed by averaging z-scores from the Keep track task and the Running span task.
Changes on the inhibition composite measure (Proximal outcome). | within the 2 weeks before intervention starts; 3rd week after intervention starts (after the 6th training session); 6th week (after the 12th training session)
  An inhibition composite score will be computed by averaging z-scores from the Anti-saccade and the Victoria Stroop Test.

SECONDARY OUTCOMES:
Transfer to complex working memory measure: the Alpha-span task (Distal outcome). | within the 2 weeks before intervention starts; 1st week after intervention starts (after the 3rd training session); 3rd week (after the 6th training session); 4th week (after the 9th training session); 6th week (after the 12th training session).
  Accuracy on the alphabetic portion of the Alpha-span task
Transfer to complex working memory measure: the Reading span task (Distal outcome). | within the 2 weeks before intervention starts; 1st week after intervention starts (after the 3rd training session); 3rd week (after the 6th training session); 4th week (after the 9th training session); 6th week (after the 12th training session).
  Accuracy on the Reading span task.
Transfer to complex working memory measure: the virtual car ride task (Distal outcome). | within the 2 weeks before intervention starts; 1st week after intervention starts (after the 3rd training session); 3rd week (after the 6th training session); 4th week (after the 9th training session); 6th week (after the 12th training session).
  Average z-score computed with the verbal and visual (accuracy and RT) components of the divided attention virtual reality task.
Brain structure: Regional gray matter volumes in Prefrontal and lateral temporal cortices, Basal ganglia and Hippocampi. | within the 2 weeks before intervention starts; 3rd week after intervention starts (after the 6th training session); 6th week (after the 12th training session)
  A T1-weighted 3D-MPRAGE sequence (TR/TE 2300/2.98ms, Fa 9°, FOV = 256*256, matrix 256*256, voxels 1mm³, 192 slices) will be used to measure regional gray matter volume.
Brain structure: Cortical thickness in Prefrontal regions and lateral temporal cortices. | within the 2 weeks before intervention starts; 3rd week after intervention starts (after the 6th training session); 6th week (after the 12th training session)
  A T1-weighted 3D-MPRAGE sequence (TR/TE 2300/2.98ms, Fa 9°, FOV = 256*256, matrix 256*256, voxels 1mm³, 192 slices) will be used to measure cortical thickness (FreeSurfer 5.3).
Brain function: Updating related activation. | within the 2 weeks before intervention starts; 3rd week after intervention starts (after the 6th training session); 6th week (after the 12th training session)
  Functional activations. Simultaneous multislice (accelerator factor = 6), echo polar (EPI) imaging: TR/TE 785/30 ms, Fa 54°, FOV 192*192, matrix 64*64, voxels 3 mm³, 39 slices) will be measured in association with a N-back task.
Brain function: Inhibition related activation. | within the 2 weeks before intervention starts; 3rd week after intervention starts (after the 6th training session); 6th week (after the 12th training session)
  Functional activations. Simultaneous multislice (accelerator factor = 6), echo polar (EPI) imaging: TR/TE 785/30 ms, Fa 54°, FOV 192*192, matrix 64*64, voxels 3 mm³, 39 slices) will be measured in association with a counting stroop.

OTHER OUTCOMES:
Effect of moderators: Polymorphisms. | 3rd week after intervention starts (after the 6th training session)
  Presence/absence of polymorphisms : Brain-derived neurotrophic factor (BDNF), Catechol-O-Methyltransferase (COMT) and Apolipoprotein (APOE)-ε4 taken from a salivary sample collected using an Oragene OG-500 collection kit.
Effect of moderators: Cognitive reserve proxies. | within the 2 weeks before intervention starts
  Scores on the reserve-proxy questionnaire (from Rami L, Valls-Pedret C, Bartres-Faz D, et al. 2011).
Effect of moderators: Intracranial volume. | within the 2 weeks before intervention starts
  Overall intracranial volume taken from MRI scan with a T1-weighted 3D-MPRAGE sequence (TR/TE 2300/2.98ms, Fa 9°, FOV = 256*256, matrix 256*256, voxels 1mm³, 192 slices).
Effect of moderators: White Matter Lesions (WML). | within the 2 weeks before intervention starts
  The WML will be quantified in mm3 (De Carli et al. 2005) from the FLAIR sequence (TR/TE 9000/120 ms, Fa 90°, FOV 240*240, matrix 256*256, voxels 0.9*0.9*3 mm, 48 slices).
Effect of moderators: Regional gray matter volumes in Prefrontal and lateral temporal cortices, Basal ganglia and Hippocampi. | within the 2 weeks before intervention starts
  A T1-weighted 3D-MPRAGE sequence (TR/TE 2300/2.98ms, Fa 9°, FOV = 256*256, matrix 256*256, voxels 1mm³, 192 slices) will be used to measure regional gray matter volume.
Effect of moderators: Cortical thickness in Prefrontal regions and lateral temporal cortices. | within the 2 weeks before intervention starts
  A T1-weighted 3D-MPRAGE sequence (TR/TE 2300/2.98ms, Fa 9°, FOV = 256*256, matrix 256*256, voxels 1mm³, 192 slices) will be used to measure cortical thickness (FreeSurfer 5.3).
Effect of moderators: Task related activation in prefrontal and lateral temporal cortices, Basal ganglia and Hippocampi. | within the 2 weeks before intervention starts
  Functional activations. Simultaneous multislice (accelerator factor = 6), echo polar (EPI) imaging: TR/TE 785/30 ms, Fa 54°, FOV 192*192, matrix 64*64, voxels 3 mm³, 39 slices) will be measured in association with a N-back task and a counting stroop.
Effect of moderators: Sex. | within the 2 weeks before intervention starts
  Male vs Female.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Belleville, PhD, Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verty LV, Mellah S, Maltezos S, Boujut A, Lussier M, Bherer L, Belleville S. Youth-like brain activation linked with greater cognitive training gains in older adults: Insights from the ACTOP study. Cortex. 2024 Jul;176:221-233. doi: 10.1016/j.cortex.2024.04.013. Epub 2024 May 17. PMID 38805784
- [Derived] Boujut A, Verty LV, Maltezos S, Lussier M, Mellah S, Bherer L, Belleville S. Effects of Computerized Updating and Inhibition Training in Older Adults: The ACTOP Three-Arm Randomized Double-Blind Controlled Trial. Front Neurol. 2020 Dec 3;11:606873. doi: 10.3389/fneur.2020.606873. eCollection 2020. PMID 33343503
- [Derived] Boujut A, Mellah S, Lussier M, Maltezos S, Verty LV, Bherer L, Belleville S. Assessing the Effect of Training on the Cognition and Brain of Older Adults: Protocol for a Three-Arm Randomized Double-Blind Controlled Trial (ACTOP). JMIR Res Protoc. 2020 Nov 24;9(11):e20430. doi: 10.2196/20430. PMID 33231556